CLINICAL TRIAL: NCT04810377
Title: Safety and Efficacy of Endoscopic Ultrasound-Guided Gastroenterostomy for the Treatment of Malignant Gastric Outlet Obstruction
Brief Title: Endoscopic Ultrasound-Guided Gastroenterostomy for Malignant Gastric Outlet Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-2020-3601-298
Record Dates: First submitted 2021-02-18; First posted 2021-03-23 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Malignant Gastric Outlet Obstruction
Keywords: EUS-Guided gastro-enterostomy; Safety; Efficacy

STUDY DESIGN:
Intervention Model Description: This is a prospective study that evaluates EUS-guided gastroenterostomy in a group of participants with diagnosis of malignant gastric outlet obstruction. Patients are sequentially recruited as diagnosed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EUS-guided gastroenterostomy in malignant gastric outlet obstruction (Experimental): The patients with malignant gastric outlet obstruction will be confirmed as follows: Histopathological report of cancer, thoracoabdominal tomography and impaired tolerance to oral feeding (tolerance to liquids only or null).
  Interventions: Procedure: EUS-guided gastroenterostomy

INTERVENTIONS:
Procedure: EUS-guided gastroenterostomy — First after an upper endoscopy is performed, a catheters passed throughout the endoscope channel and with x-ray verification, a guide wire is passed up to the third portion of duodenal loop. then small intestinal is filled with saline solution up to 1500cc and contrast solution. Then an endoscopic ultrasound examination will be carried out where a loop of the small intestine that is located less than 2 cm apart from the gastric wall will be looked for. Once the intestinal loop is identified a direct antegrade puncture will be performed with a luminal apposition prosthesis release system . Finally, correct position is verified with x-ray and we will look for any misplacement or leakage during this process or the presence of bleeding. Endoscopic treatment will be performed if necessary. Subsequently, the participants will go to monthly follow-up with clinical evaluation, laboratory and radiological test will be carried out until the participants dies.

SUMMARY:
Malignant gastric outlet obstruction is a very disabling complication of patients with gastric, duodenal, ampullary, pancreatic, or bile duct cancer and worsens their prognosis. Current treatments have reported a similar complication rate and higher mortality in surgically treated patients. Recently, the creation of endoscopic ultrasound-guided gastroenterostomy (EUS) has shown promising results in these patients. The aim of this research is to determine the safety and efficacy of EUS-guided gastro-enterostomy in the treatment of patients with malignant gastric outlet obstruction.

DETAILED DESCRIPTION:
Malignant gastric outlet obstruction is a very disabling complication that occurs in 15% to 25% of patients with gastric, duodenal, ampullary, pancreatic, or bile duct cancer and worsens their prognosis. Roux-en-Y gastrojejunostomy is considered the gold standard treatment with technical success of 98.6% (97-3% -99.9%) and clinical success of 80.1% with patency of 169.2 (136.8-201.7) days. On the other hand, the technical success reported for self-expanding metal stents is 96.2% (94.1% vs. 98.4%), technical success is 79.4%, and patency at 6 months was only 57%. However, complications occur in a similar way in both forms of treatment (major complications in 6% and late complications in 17% in both, but mortality is higher in the group treated with Roux-en-Y gastrojejunostomy (29% vs. 17%). , p <0.001) Recently, the creation of endoscopic ultrasound-guided gastroenterostomy has shown success rates of over 90% in case series, but prospective studies evaluating the safety and efficacy of the procedure are lacking. The aim of this research to determine the safety and efficacy of EUS-guided gastro-enterostomy in the treatment of patients with malignant gastric outlet obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders over 18 years of age with gastric outlet obstruction syndrome secondary to stage III or more at gastric, duodenal or pancreatic cancer who are candidates for palliative treatment, who do not want surgical treatment.

  * Diagnosis confirmed as follows:

    * Histopathological report of cancer.
    * Simple and contrasted thoracoabdominal tomography.
    * Tolerance to oral feeding based on liquids only or null.

Exclusion Criteria:

* Patients who do not accept the signing of the informed consent.

  * Postoperative patients with Roux-en-Y gastrojejunostomy.
  * Patients with large volume ascites.
  * Patients with malignant obstruction distal to the jejunal puncture.
  * Pregnant women.
  * Patients with a Karnofsky index less than 50 or an E.C.O.G. greater than or equal to 4 points.
  * Patients in whom any endoscopic procedure has been contraindicated for any reason.
  * Patients who want to undergo surgical treatment as an initial option.
  * Patients with malignant biliary obstruction without endoscopic treatment at the time of gastric outflow tract obstruction presentation.

Elimination Criteria:

* Patients who undergo the endoscopic procedure but cannot be completed due to transmural invasion of malignancy, hemorrhage or inability to puncture the intestinal loop with any method described, puncture site> 2cm away from the gastric wall or inability to pass the guidewire through obstruction (unless direct technique is performed).
* Patients who do not attend follow-up.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Incidence of immediate adverse events in patients with gastric outflow tract obstruction treated by EUS-guided gastro-enterostomy. | Adverse events will be recorded during the first 24 hours of the procedure
  To evaluate the proportion of patients that presents with bleeding , prostheses misplacement or perforation.
Incidence of early-term adverse events in patients with gastric outflow tract obstruction treated by EUS-guided gastro-enterostomy. | Adverse events will be recorded after the first day up to 30 days of the procedure
  we will record the proportion of patients that presents with migration, clogging, stenosis at gastro-enterostomy site or leakage.
Incidence of mid-term adverse events in patients with gastric outflow tract obstruction treated by EUS-guided gastro-enterostomy. | Adverse events will be recorded from the first month up to the third month after procedure
  we will record the proportion of patients that presents with migration, clogging, stenosis at gastro-enterostomy site or leakage.
Incidence of long-term adverse events in patients with gastric outflow tract obstruction treated by EUS-guided gastro-enterostomy. | Adverse events will be recorded after the third month of the stent placement up to study completion, an average of 6 months
  we will record the proportion of patients that presents with migration, clogging, stenosis at gastro-enterostomy site or leakage.
Incidence of the correct stent placement for endoscopic ultrasound gastro-enterostomy anastomosis creation at the desired loop | During each procedure correct stent placement will be assessed
  Technical success: We will determine the ability to place the stents in the desired loop and in a correct position.

SECONDARY OUTCOMES:
Improvement in tolerance to oral feeding assessed by the gastric outlet obstruction scoring system (GOOSS) in patients with gastric outflow tract obstruction treated by EUS-guided gastro-enterostomy | Immediately after the intervention/procedure/surgery and every month through study completion, an average of 6 months
  Clinical success: Defined as an increase in tolerance to oral feeding, assessed by GOOSS: 0 = no/inadequate oral intake, 1 = liquids/thickened liquids, 2 = semisolids/low residue diet, 3 = unmodified diet. A higher score means a better outcome.
Changes in quality of life assessed by the self-report health-related quality of life questionnaire in patients with gastric outflow tract obstruction treated by EUS-guided gastro-enterostomy. | Baseline and every month after the intervention/procedure/surgery through study completion, an average of 6 months.
  Quality of life will be measured with the short form survey (SF-36 questionnaire). It consists of physical and mental component scores ranging from 0 to 100; a higher scores means a better outcome, a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Changes of functional impairment assessed by Karnofsky Performance Scale Index in patients with gastric outflow tract obstruction treated by EUS-guided gastro-enterostomy. | Baseline and every month after the intervention/procedure/surgery through study completion, an average of 6 months.
  The Karnofsky Performance Scale Index allows patients to be classified as to their functional impairment. The lower scores means worst prognosis: 100-80 means that the patient is able to perform normal activities; 70-50 points means that the patient is unable to work; able to live at home and care for most personal needs, and 40-0 points means that the patient is unable to care for self; requires equivalent of hospital care and disease may be progressing rapidly.
Changes in functional status with Eastern Cooperative Oncology Group (ECOG) performance scale in patients with gastric outflow tract obstruction treated by EUS-guided gastro-enterostomy. | Baseline and every month after the intervention/procedure/surgery through study completion, an average of 6 months.
  The ECOG Scale of performance status describes patients functionality. Lower points means best outcomes.0: fully active. 1: Restricted in some physical activities. 2: Capable of all self-care but unable to carry our any work activities, more than 50% of walking hours. 3: limited self-care, confined to bed or chair more tan 50% of walking hours. 4: Completely disabled. Totally confined to bed or chair. 5: Dead.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar V Hernández Mondragón, MD, Principal Investigator — IMSS
Locations (1):
- Centro Medico Nacional Siglo XXI Hospital de Especialidades, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suder-Castro LS, Ramirez-Solis ME, Hernandez-Guerrero AI, de la Mora-Levy JG, Alonso-Larraga JO, Hernandez-Lara AH. Predictors of self-expanding metallic stent dysfunction in malignant gastric outlet obstruction. Rev Gastroenterol Mex (Engl Ed). 2020 Jul-Sep;85(3):275-281. doi: 10.1016/j.rgmx.2019.07.009. Epub 2020 Mar 27. English, Spanish. PMID 32229056
- [Background] Lundstrom B, Fagerberg G. Clinical problems in relation to breast cancer screening with mammography. A preliminary report. Acta Chir Scand Suppl. 1984;519:61-3. PMID 6595925
- [Background] Metges PJ, Cosnard G, Pailler JL, Chantome M, Flageat J. [Trapped popliteal artery. Early diagnosis by dynamic tests during arteriography (author's transl)]. J Radiol. 1981 May;62(5):331-3. French. PMID 7288729
- [Background] Storm AC, Ryou M. Advances in the endoscopic management of gastric outflow disorders. Curr Opin Gastroenterol. 2017 Nov;33(6):455-460. doi: 10.1097/MOG.0000000000000403. PMID 28984645
- [Background] Laasch HU, Martin DF, Maetani I. Enteral stents in the gastric outlet and duodenum. Endoscopy. 2005 Jan;37(1):74-81. doi: 10.1055/s-2004-826103. No abstract available. PMID 15657863
- [Background] Balderramo DC. [Gastric outlet obstruction]. Rev Esp Enferm Dig. 2008 Feb;100(2):98-9. doi: 10.4321/s1130-01082008000200007. No abstract available. Spanish. PMID 18366268
- [Background] Chandrasegaram MD, Eslick GD, Mansfield CO, Liem H, Richardson M, Ahmed S, Cox MR. Endoscopic stenting versus operative gastrojejunostomy for malignant gastric outlet obstruction. Surg Endosc. 2012 Feb;26(2):323-9. doi: 10.1007/s00464-011-1870-3. Epub 2011 Sep 5. PMID 21898024
- [Background] Jeurnink SM, Steyerberg EW, van Hooft JE, van Eijck CH, Schwartz MP, Vleggaar FP, Kuipers EJ, Siersema PD; Dutch SUSTENT Study Group. Surgical gastrojejunostomy or endoscopic stent placement for the palliation of malignant gastric outlet obstruction (SUSTENT study): a multicenter randomized trial. Gastrointest Endosc. 2010 Mar;71(3):490-9. doi: 10.1016/j.gie.2009.09.042. Epub 2009 Dec 8. PMID 20003966
- [Background] Beltcheva I, Stoytchev T. Central depressive action of two N-aminomethyl derivatives of diethylpyridinedione. Acta Physiol Pharmacol Bulg. 1983;9(1):35-43. PMID 6684873
- [Background] Ucar K. The effects of histamine H2 receptor antagonists on melanogenesis and cellular proliferation in melanoma cells in culture. Biochem Biophys Res Commun. 1991 May 31;177(1):545-50. doi: 10.1016/0006-291x(91)92018-f. PMID 1904222
- [Background] Espinel J, Vivas S, Munoz F, Jorquera F, Olcoz JL. Palliative treatment of malignant obstruction of gastric outlet using an endoscopically placed enteral Wallstent. Dig Dis Sci. 2001 Nov;46(11):2322-4. doi: 10.1023/a:1012378509762. PMID 11713929
- [Background] Phillips MS, Gosain S, Bonatti H, Friel CM, Ellen K, Northup PG, Kahaleh M. Enteral stents for malignancy: a report of 46 consecutive cases over 10 years, with critical review of complications. J Gastrointest Surg. 2008 Nov;12(11):2045-50. doi: 10.1007/s11605-008-0598-4. Epub 2008 Jul 22. PMID 18648893
- [Background] Meylan J, Schindler AM, Kaji T. [Hormonal balance in 2 cases of testicular feminization]. Gynakol Rundsch. 1973;13:Suppl 1:66-7. No abstract available. French. PMID 4798937
- [Background] Jang S, Stevens T, Lopez R, Bhatt A, Vargo JJ. Superiority of Gastrojejunostomy Over Endoscopic Stenting for Palliation of Malignant Gastric Outlet Obstruction. Clin Gastroenterol Hepatol. 2019 Jun;17(7):1295-1302.e1. doi: 10.1016/j.cgh.2018.10.042. Epub 2018 Oct 31. PMID 30391433
- [Background] Adler DG, Baron TH. Endoscopic palliation of malignant gastric outlet obstruction using self-expanding metal stents: experience in 36 patients. Am J Gastroenterol. 2002 Jan;97(1):72-8. doi: 10.1111/j.1572-0241.2002.05423.x. PMID 11808972
- [Background] Dormann A, Meisner S, Verin N, Wenk Lang A. Self-expanding metal stents for gastroduodenal malignancies: systematic review of their clinical effectiveness. Endoscopy. 2004 Jun;36(6):543-50. doi: 10.1055/s-2004-814434. PMID 15202052
- [Background] van Hooft JE, Dijkgraaf MG, Timmer R, Siersema PD, Fockens P. Independent predictors of survival in patients with incurable malignant gastric outlet obstruction: a multicenter prospective observational study. Scand J Gastroenterol. 2010 Oct;45(10):1217-22. doi: 10.3109/00365521.2010.487916. PMID 20459356
- [Background] Staub J, Siddiqui A, Taylor LJ, Loren D, Kowalski T, Adler DG. ERCP performed through previously placed duodenal stents: a multicenter retrospective study of outcomes and adverse events. Gastrointest Endosc. 2018 Jun;87(6):1499-1504. doi: 10.1016/j.gie.2018.01.040. Epub 2018 Feb 6. PMID 29425886
- [Background] Mutignani M, Tringali A, Shah SG, Perri V, Familiari P, Iacopini F, Spada C, Costamagna G. Combined endoscopic stent insertion in malignant biliary and duodenal obstruction. Endoscopy. 2007 May;39(5):440-7. doi: 10.1055/s-2007-966327. PMID 17516351
- [Background] Ruggiero J, Manzini G, Quadrifoglio F. Ionic and nonionic contributions to the free-energy change in the B-Z transition of alternating polydeoxynucleotides in aqueous solution. Biopolymers. 1987 Nov;26(11):1975-9. doi: 10.1002/bip.360261112. No abstract available. PMID 3689879
- [Background] Kim CG, Choi IJ, Lee JY, Cho SJ, Park SR, Lee JH, Ryu KW, Kim YW, Park YI. Covered versus uncovered self-expandable metallic stents for palliation of malignant pyloric obstruction in gastric cancer patients: a randomized, prospective study. Gastrointest Endosc. 2010 Jul;72(1):25-32. doi: 10.1016/j.gie.2010.01.039. Epub 2010 Apr 9. PMID 20381802
- [Background] Kim JH, Song HY, Shin JH, Choi E, Kim TW, Jung HY, Lee GH, Lee SK, Kim MH, Ryu MH, Kang YK, Kim BS, Yook JH. Metallic stent placement in the palliative treatment of malignant gastroduodenal obstructions: prospective evaluation of results and factors influencing outcome in 213 patients. Gastrointest Endosc. 2007 Aug;66(2):256-64. doi: 10.1016/j.gie.2006.12.017. PMID 17643698
- [Background] Jang JK, Song HY, Kim JH, Song M, Park JH, Kim EY. Tumor overgrowth after expandable metallic stent placement: experience in 583 patients with malignant gastroduodenal obstruction. AJR Am J Roentgenol. 2011 Jun;196(6):W831-6. doi: 10.2214/AJR.10.5861. PMID 21606277
- [Background] Sasaki T, Isayama H, Nakai Y, Takahara N, Hamada T, Mizuno S, Mohri D, Yagioka H, Kogure H, Arizumi T, Togawa O, Matsubara S, Ito Y, Yamamoto N, Sasahira N, Hirano K, Toda N, Tada M, Koike K. Clinical outcomes of secondary gastroduodenal self-expandable metallic stent placement by stent-in-stent technique for malignant gastric outlet obstruction. Dig Endosc. 2015 Jan;27(1):37-43. doi: 10.1111/den.12321. Epub 2014 Aug 28. PMID 24995858
- [Background] Ly J, O'Grady G, Mittal A, Plank L, Windsor JA. A systematic review of methods to palliate malignant gastric outlet obstruction. Surg Endosc. 2010 Feb;24(2):290-7. doi: 10.1007/s00464-009-0577-1. Epub 2009 Jun 24. PMID 19551436
- [Background] Mehta S, Hindmarsh A, Cheong E, Cockburn J, Saada J, Tighe R, Lewis MP, Rhodes M. Prospective randomized trial of laparoscopic gastrojejunostomy versus duodenal stenting for malignant gastric outflow obstruction. Surg Endosc. 2006 Feb;20(2):239-42. doi: 10.1007/s00464-005-0130-9. Epub 2005 Dec 9. PMID 16362479
- [Background] Yamao K, Kitano M, Kayahara T, Ishida E, Yamamoto H, Minaga K, Yamashita Y, Nakajima J, Asada M, Okabe Y, Osaki Y, Chiba Y, Imai H, Kudo M. Factors predicting through-the-scope gastroduodenal stenting outcomes in patients with gastric outlet obstruction: a large multicenter retrospective study in West Japan. Gastrointest Endosc. 2016 Nov;84(5):757-763.e6. doi: 10.1016/j.gie.2016.03.1498. Epub 2016 Apr 4. PMID 27055762
- [Background] Hori Y, Naitoh I, Hayashi K, Ban T, Natsume M, Okumura F, Nakazawa T, Takada H, Hirano A, Jinno N, Togawa S, Ando T, Kataoka H, Joh T. Predictors of outcomes in patients undergoing covered and uncovered self-expandable metal stent placement for malignant gastric outlet obstruction: a multicenter study. Gastrointest Endosc. 2017 Feb;85(2):340-348.e1. doi: 10.1016/j.gie.2016.07.048. Epub 2016 Jul 27. PMID 27475489
- [Background] Sato T, Hara K, Mizuno N, Hijioka S, Imaoka H, Niwa Y, Tajika M, Tanaka T, Ishihara M, Shimizu Y, Bhatia V, Kobayashi N, Endo I, Maeda S, Nakajima A, Kubota K, Yamao K. Gastroduodenal stenting with Niti-S stent: long-term benefits and additional stent intervention. Dig Endosc. 2015 Jan;27(1):121-9. doi: 10.1111/den.12300. Epub 2014 Apr 22. PMID 24754262
- [Background] Fritscher-Ravens A, Mosse CA, Mills TN, Mukherjee D, Park PO, Swain P. A through-the-scope device for suturing and tissue approximation under EUS control. Gastrointest Endosc. 2002 Nov;56(5):737-42. doi: 10.1067/mge.2002.129084. PMID 12397289
- [Background] Fritscher-Ravens A, Mosse CA, Mukherjee D, Mills T, Park PO, Swain CP. Transluminal endosurgery: single lumen access anastomotic device for flexible endoscopy. Gastrointest Endosc. 2003 Oct;58(4):585-91. doi: 10.1016/s0016-5107(03)02006-6. PMID 14520300
- [Background] Binmoeller KF, Shah JN. Endoscopic ultrasound-guided gastroenterostomy using novel tools designed for transluminal therapy: a porcine study. Endoscopy. 2012 May;44(5):499-503. doi: 10.1055/s-0032-1309382. Epub 2012 Apr 24. PMID 22531985
- [Background] Amin S, Sethi A. Endoscopic Ultrasound-Guided Gastrojejunostomy. Gastrointest Endosc Clin N Am. 2017 Oct;27(4):707-713. doi: 10.1016/j.giec.2017.06.009. PMID 28918806
- [Background] Irani S, Baron TH, Itoi T, Khashab MA. Endoscopic gastroenterostomy: techniques and review. Curr Opin Gastroenterol. 2017 Sep;33(5):320-329. doi: 10.1097/MOG.0000000000000389. PMID 28767501
- [Background] Itoi T, Itokawa F, Uraoka T, Gotoda T, Horii J, Goto O, Moriyasu F, Moon JH, Kitagawa Y, Yahagi N. Novel EUS-guided gastrojejunostomy technique using a new double-balloon enteric tube and lumen-apposing metal stent (with videos). Gastrointest Endosc. 2013 Dec;78(6):934-939. doi: 10.1016/j.gie.2013.09.025. PMID 24237949
- [Background] Itoi T, Ishii K, Tanaka R, Umeda J, Tonozuka R. Current status and perspective of endoscopic ultrasonography-guided gastrojejunostomy: endoscopic ultrasonography-guided double-balloon-occluded gastrojejunostomy (with videos). J Hepatobiliary Pancreat Sci. 2015 Jan;22(1):3-11. doi: 10.1002/jhbp.148. Epub 2014 Aug 24. PMID 25155270
- [Background] Itoi T, Ishii K, Ikeuchi N, Sofuni A, Gotoda T, Moriyasu F, Dhir V, Teoh AY, Binmoeller KF. Prospective evaluation of endoscopic ultrasonography-guided double-balloon-occluded gastrojejunostomy bypass (EPASS) for malignant gastric outlet obstruction. Gut. 2016 Feb;65(2):193-5. doi: 10.1136/gutjnl-2015-310348. Epub 2015 Aug 17. No abstract available. PMID 26282674
- [Background] Anastosatu C, Dutu S. [Contribution of pulmonary function tests to pneumonology. Report]. Ftiziologia. 1973 Jan-Feb;22(1):1-8. No abstract available. Romanian. PMID 4690188
- [Background] Fan W, Tan S, Wang J, Wang C, Xu H, Zhang L, Liu L, Fan Z, Tang X. Clinical outcomes of endoscopic ultrasound-guided gastroenterostomy for gastric outlet obstruction: a systematic review and meta-analysis. Minim Invasive Ther Allied Technol. 2022 Feb;31(2):159-167. doi: 10.1080/13645706.2020.1792500. Epub 2020 Jul 16. PMID 32672479
- [Background] Barthet M, Binmoeller KF, Vanbiervliet G, Gonzalez JM, Baron TH, Berdah S. Natural orifice transluminal endoscopic surgery gastroenterostomy with a biflanged lumen-apposing stent: first clinical experience (with videos). Gastrointest Endosc. 2015 Jan;81(1):215-8. doi: 10.1016/j.gie.2014.09.039. PMID 25527056